CLINICAL TRIAL: NCT01839253
Title: The Effect of Antihypertensive Agents Concerning With Hemodynamics and Reduction of Anaesthetics in Orthognathic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4-2012-0422
Record Dates: First submitted 2013-04-17; First posted 2013-04-24 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Orthognathic Surgery
Keywords: antihypertensive agents; hemodynamic; anesthetics reduction; orthognathic surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Atenolol (Experimental): In each group, premedication with either b-blocker (Atenolol) or ACE inhibitor (enalapril) or nothing (control group) in the preparation room.
  Interventions: Drug: b-blocker(Atenolol)
- Enalapril (Active Comparator): In each group, premedication with either b-blocker (Atenolol) or ACE inhibitor (enalapril) or nothing (control group) in the preparation room.
  Interventions: Drug: ACE inhibitor(Enapril)
- control (Placebo Comparator): none of antihypertensive agents
  Interventions: Other: control

INTERVENTIONS:
Drug: b-blocker(Atenolol)
  Arms: Atenolol
Drug: ACE inhibitor(Enapril)
  Arms: Enalapril
Other: control
  Arms: control

SUMMARY:
For those who receive hypotensive anesthesia in orthognathic surgeries, the investigators premedicate with anti-hypertensive agent so that it decreases the occurence of tachycardia and the rebound hypertension due to hypotensive anesthesia, enabling us to compare hemodynamic stability and reduction of anesthetic agents during the operation.

ELIGIBILITY:
Inclusion Criteria:

1. ASA class I-II
2. obtaining written informed consent from the parents
3. aged 18-29 years who were undergoing orthognathic surgery.

Exclusion Criteria:

1. Hypertension patients with anti-hypertensive agents
2. chronic renal failure or End stage renal disease patients.
3. renal artery stenosis history.
4. Patients who are with medication due to systemic disease.
5. symptomatic asthma
6. Drug hyperactivity
7. neurological or psychiatric illnesses
8. mental retardation
9. patients who can't read the consent form due to illiterate or foreigner

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2012-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
the influence of antihypertensive agents on hemodynamic stability | From the beginning until the end of hypoetensive anesthesiaan expected average of 65 mins.(From manipulration of Mandible to maxilla)
  Total minutes when the MAP is lower than 55mmHg and higher than 65mmHg (min) , The time below 55 mmHg(min) , The total time above 65 mmHg (min) Total remifentanil amount, total NTG amount, total phenylephrine amount Arterial gas analysis 4 times after induction, at the start of manipulation of mandible, at the start of manipulation of maxilla, at the end of surgery.
  Pr-operative and post-operative lab (Hb, Bun, Cr, OT, PT, Na, K) Intraoperative total fluid, total urine amount, total blood loss, transfusion amount.

SECONDARY OUTCOMES:
reduction of anaesthetics with control | From the beginning until the end of hypoetensive anesthesia an expected average of 65 mins.(From manipulration of Mandible to maxilla)
  Total minutes when the MAP is lower than 55mmHg and higher than 65mmHg (min) , The time below 55 mmHg(min) , The total time above 65 mmHg (min) Total remifentanil amount, total NTG amount, total phenylephrine amount Arterial gas analysis 4 times after induction, at the start of manipulation of mandible, at the start of manipulation of maxilla, at the end of surgery.
  Pr-operative and post-operative lab (Hb, Bun, Cr, OT, PT, Na, K) Intraoperative total fluid, total urine amount, total blood loss, transfusion amount.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, Seoul, South Korea